CLINICAL TRIAL: NCT01242176
Title: Relative Bioavailability of 25 mg BI 10773 (Final Formulation) Compared to 25 mg BI 10773 XX (Trial Formulation 2) Following Oral Administration in Healthy Male and Female Volunteers (an Open-label, Randomised, Single-dose, Two-way Crossover Study)
Brief Title: Relative Bioavailability of Empagliflozin (BI 10773) (Final Formulation) Compared to Empagliflozin (BI 10773 XX) (Trial Formulation 2) in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.51; 2010-022469-81 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-11-10; First posted 2010-11-16 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin

ARMS (2):
- BI 10773 Final Formulation (Experimental): one single film-coated tablet in the morning
  Interventions: Drug: BI 10773 (Final Formulation)
- BI 10773 XX Trial Formulation 2 (Experimental): one single dose tablet in the morning
  Interventions: Drug: BI 10773 XX (Trial Formulation 2)

INTERVENTIONS:
Drug: BI 10773 XX (Trial Formulation 2) — one single dose tablet in the morning
  Arms: BI 10773 XX Trial Formulation 2
Drug: BI 10773 (Final Formulation) — one single film-coated tablet in the morning
  Arms: BI 10773 Final Formulation

SUMMARY:
The objective of the study is to investigate the relative bioavailability of the final tablet formulation (FF) of BI 10773 in comparison to the tablet formulation 2 (TF2).

ELIGIBILITY:
Inclusion criteria:

Healthy male and female subjects

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.51.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Empa FF / Empa TF2: Single dose of 25mg of empagliflozin (empa) final formulation (FF) followed by a single dose of 25mg empa trial formulation 2 (TF2), with a washout period of at least 7 days between treatments.
- Empa TF2 / Empa FF: Single dose of 25mg empagliflozin (empa) trial formulation 2 (TF2) followed by a single dose of 25mg of empa final formulation (FF), with a washout period of at least 7 days between treatments.
Period: First Intervention
Arm/Group | Empa FF / Empa TF2 | Empa TF2 / Empa FF
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Empa FF / Empa TF2 | Empa TF2 / Empa FF
Started | 12 | 12
Completed | 11 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Non-compliant with protocol | 1 | 0
Period: Second Intervention
Arm/Group | Empa FF / Empa TF2 | Empa TF2 / Empa FF
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Overall: An open-label, randomised, two-way crossover study. The two treatments administered were
  * A single dose of empagliflozin (empa) 25mg, final formulation
  * A single dose of empa 25mg, trial formulation 2
  Between drug administrations there was a washout period of at least 7 days.
Arm/Group | Study Overall
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 extrapolated to infinity.
  Note the standard deviation is actually the coefficient of variation (CV (%)).
Time Frame: 30 minutes (mins) before drug administration and 20min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h after drug administration
Population: Pharmacokinetic (PK) set included all subjects who took at least one dose of study medication and who provided evaluable data for at least one observation for at least one primary PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Mean (Standard Deviation); unit: nmol*h/L
Groups:
- Empa FF: Single dose of empagliflozin (empa) 25 mg, final formulation (FF), following an overnight fast of at least 10 hours.
- Empa TF2: Single dose of empagliflozin (empa) 25 mg, trial formulation 2 (TF2), following an overnight fast of at least 10 hours.
Arm/Group | Empa FF | Empa TF2
Number analyzed (Participants) | 21 | 23
nmol*h/L | 5200 (20.7) | 5090 (17.7)
Statistical Analysis 1: Comparison: Empa FF vs Empa TF2; Ratio calculated as empa final formulation divided by empa trial formulation 2; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 101.67, 90% CI 2-sided [98.10 to 105.37], Standard Deviation 6.7 — Standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of empagliflozin (empa) in plasma.
  Note the standard deviation is actually the CV (%).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Empa FF | Empa TF2
Number analyzed (Participants) | 21 | 23
nmol/L | 764 (26.5) | 764 (23.0)
Statistical Analysis 1: Comparison: Empa FF vs Empa TF2; Ratio calculated as empa final formulation divided by empa trial formulation 2; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 99.46, 90% CI 2-sided [90.18 to 109.68], Standard Deviation 18.7 — Standard deviation is actually the gCV

3. Secondary Outcome: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 to the time of the last quantifiable data point.
  Note the standard deviation is actually the CV (%).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Empa FF | Empa TF2
Number analyzed (Participants) | 21 | 23
nmol*h/L | 5140 (20.8) | 5030 (18.0)
Statistical Analysis 1: Comparison: Empa FF vs Empa TF2; Ratio calculated as empa final formulation divided by empa trial formulation 2; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 101.80, 90% CI 2-sided [98.26 to 105.48], Standard Deviation 6.7 — Standard deviation is actually the gCV

ADVERSE EVENTS:
Time Frame: From drug administration until end of study visit, up to 10 days
Arm/Group | Empa FF | Empa TF2
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/23
Other Adverse Events (participants affected / at risk) | 1/22 | 4/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empa FF (N=22) | Empa TF2 (N=23)
Migraine with aura (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa FF (N=22) | Empa TF2 (N=23)
Headache (Nervous system disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes